CLINICAL TRIAL: NCT06554652
Title: Tracer Navigated Selective Neck Dissection Versus Modified Neck Dissection in Papillary Thyroid Cancer With Limited Lymph Node Metastasis in the Lateral Neck: A Randomized, Noninferiority Phase III Trial
Brief Title: Selective Neck Dissection Versus Modified Neck Dissection in PTC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yu Wang, Chief of Head and Neck Surgery, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SELECTION
Record Dates: First submitted 2024-07-27; First posted 2024-08-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-05

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Selective neck dissection (Experimental)
  Interventions: Procedure: Lymph node tracer navigated selective neck dissection
- Modified neck dissection (Active Comparator)
  Interventions: Procedure: Modified neck dissection

INTERVENTIONS:
Procedure: Lymph node tracer navigated selective neck dissection — Selective lateral lymph node dissection (after injection of tracer, lymph nodes in compartment III-IV are dissected; if there is dyed lymph node in compartment IIA, then IIA is dissected).
  Arms: Selective neck dissection
Procedure: Modified neck dissection — Lymph nodes in compartment IIA, IIB, III, IV, VB are dissected.
  Arms: Modified neck dissection

SUMMARY:
This study is a phase III, randomized controlled, open label non inferiority study. Patients who meet the inclusion criteria are randomly assigned 1:1 to either the experimental group (selective neck dissection) or the control group (modified neck dissection), with LRFS as the primary endpoint. The aim of the study is to evaluate the safety of selective neck dissection in papillary carcinoma with limited number of lymph node metastases in the lateral neck, and the quality of life compared with modified neck dissection.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed PTC;
* Age range: 14-80 years old;
* Preoperative fine needle aspiration confirms lymph node metastasis in the lateral neck
* Ultrasound and CT suggest that metastatic/suspected metastatic lymph nodes are limited to compartment IV, with 1-2 lymph node metastases and <1cm in short diameter. The lymph nodes have no central necrosis, liquefaction, peripheral enhancement, or disappearance of adjacent fat spaces (predicting unobstructed lymphatic vessels);
* Thyroid tumors without extra thyroidal extension;
* Enough thyroid volume to inject tracer.

Exclusion Criteria:

* Previous neck surgery;
* Bilateral neck lymph node dissection;
* Distant metastases;
* High risk pathological subtypes or the presence of other high-risk factors for recurrence;
* Previous treatment for thyroid cancer other than endocrine therapy;
* The patient is unable to cooperate with follow-up.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Local-regional Recurrence Free Survival，LRFS | 5 years
  The time from surgery to the recurrence based on RECIST 1.1,. The definition of local-regional areas includes thyroid area, cervical I-VII lymph nodes, and retropharyngeal lymph nodes.

SECONDARY OUTCOMES:
Local-regional Recurrence Rate，LRR | 5 years
  The percentage of patients with local-regional recurrence in the total number of patients.
Progression Free Survival，PFS | 5 years
  The time from surgery to tumor progression, including local-regional recurrence and distant metastasis.
Overall Survival，OS | 5 years
  The time from surgery to patient death
Adverse Events，AE | 5 years
  The name of AE (based on NCI-CTCAE V5.0 criteria), severity, duration, and correlation with surgery.
Quality of Life as assessed by UW-QOL V4.1 | 5 years
  Quality of life assessments will be conducted at 1 week, 3 months, 1 year, 2 years, and 5 years after surgery. The QoL evaluation scale adopts the Washington University Quality of Life Questionnaire V4.1 (UW-QOL V4.1).
Quality of Life as assessed by QoL/Thyroid | 5 years
  Quality of life assessments will be conducted at 1 week, 3 months, 1 year, 2 years, and 5 years after surgery. The QoL evaluation scale adopts the Thyroid Cancer Quality of Life Scale QoL/Thyroid.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Univeristy Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided